CLINICAL TRIAL: NCT01769846
Title: The Impact of Early Mobilization Protocol in Patients in the ICU of the University Hospital of Santa Maria.
Brief Title: The Impact of Early Mobilization Protocol in Patients in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Isabella Martins de Albuquerque, Professor DSc., Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07201712.8.0000.5346
Record Dates: First submitted 2013-01-11; First posted 2013-01-17 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Muscle Weakness; Quality of Life; Weaning Acceleration; ICU Length of Stay; Muscle Thickness of the Quadriceps Femoris
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Mobilization protocol (Experimental): Early Mobilization protocol: Patients in the treatment group additionally received a progressive cycling exercise session 7 days a week, until the last day of ICU stay, using a bedside cycle ergometer (MOTOmed Letto 2, RECK-Technik GmbH & Co. KG, Betzenweiler, Germany). Cycling exercise will be realized during 30 consecutive minutes, initially in continuos and passive (classified patients with RASS - 4) exercise, at a fixed pedaling rate of 20 cycles/min and after in actively (classified patients with RASS 0), with an exercise intensity of 3-5 on the Borg rate of perceived exertion scale.
  Interventions: Other: Early mobilization protocol
- Control group (No Intervention): Group will undergo usual mobilization per standard ICU care. Conventional physical and respiratory therapy were provided by the ICU physical therapists twice daily, for approximately 30 min, 7 days per week. The protocol included vibrocompression maneuvers; lung hyperinflation by the mechanical ventilator; and tracheal aspiration, when necessary; as well as passive and active-assisted motor exercises for arms and legs, depending on the clinical course of patients.

INTERVENTIONS:
Other: Early mobilization protocol — Patients in the treatment group additionally received a cycling exercise session 7 days a week, using a bedside cycle ergometer (MOTOmed Letto 2, RECK-Technik GmbH & Co. KG, Betzenweiler, Germany). The device offers the possibility to conduct passive or active cycling at six levels of increasing resistance. The aim of each session was to have the patient cycle for 30 mins at an individually adjusted intensity level. Patients were placed in a comfortable position in between the supine and the semirecumbent position.
  Arms: Early Mobilization protocol

SUMMARY:
Advances in intensive care and mechanical ventilation (MV) in the past two decades have increased critically ill patient survival. However, some patients require prolonged MV (PMV) and are deconditioned due to respiratory insufficiency caused by underlying disease, adverse effects of medications, and prolonged immobilization. Patients in the intensive care unit (ICU) are often confined to their beds, which results in inactivity, immobility, and severe osteomyoarticular system dysfunction. Our hypothesis is that an early mobilization protocol improves muscle thickness (MT) of the quadriceps femoris, peripheral muscle strength, perceived functional status, gait speed, quality of life, duration of mechanical ventilation, ICU length of stay of the critically ill patient.

The purpose of this study is to evaluate the effects of implementation an early mobilization protocol in critically ill patients in the Intensive Care Unit of the University Hospital of Santa Maria.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or greater)
* Patients in the first 24 hours of mechanical ventilation.
* Patients in the deep sedation will be evaluated by the Richmond Agitation-Sedation Scale (score -4).
* Hemodynamically stable.

Exclusion Criteria:

* Rapidly developing neuromuscular disease
* Evolution of brain death
* Cardiopulmonary arrest
* Elevated intracranial pressure
* Ruptured/leaking aortic aneurysm
* Acute MI before peak troponin has been reached
* Absent lower limb
* Pregnancy
* Unstable fractures contributing to likely immobility
* Hospitalization prior to ICU admission >5 days
* Enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Muscle thickness (MT) of the quadriceps femoris. | Change from baseline at 14 day of ICU admission, an average of 1 month.
  MT of the quadriceps femoris will be assessed by ultrasonography (baseline and 14 day).
Muscle thickness (MT) of the diaphragm. | Change from baseline at 14 day of ICU admission, an average of 1 month.
  MT of the diaphragm will be assessed by ultrasonography (baseline and 14 day).

SECONDARY OUTCOMES:
Rectus femoris cross-sectional area | Change from baseline at 14 day of ICU admission, an average of 1 month.
  Rectus femoris cross-sectional area will be assessed by ultrasonography (baseline and 14 day).
Vastus intermedius, rectus femoris and diaphragm echo intensity. | Change from baseline at 14 day of ICU admission, an average of 1 month.
  Vastus intermedius, rectus femoris and diaphragm echo intensity will be assessed by ultrasonography (baseline and 14 day)
Rectus femoris and vastus intermedius thickness. | Change from baseline at 14 day of ICU admission, an average of 1 month.
  Rectus femoris and vastus intermedius thickness will be assessed by ultrasonography (baseline and 14 day).
Muscle strength | First day of the patient was cooperative and responsive and at day 14 of ICU admission, an average of 1 month.
  Muscle strength in arms and legs will be measured by the Medical Research Council (MRC) scale.
Gait speed | Study completion, an average of 2 months (hospital discharge)
  Gait speed will be measured by the six-meter gait speed test (GST)
Peripheral muscle strength of the lower limbs | Study completion, an average of 2 months (hospital discharge)
  Peripheral muscle strength of the lower limbs will be measured by 30 second chair stand test
Quality of life following hospital discharge | Three months after hospital discharge SF36
  Quality of life will be measured by a questionnaire 36-item Short Form Health Survey
Mortality | Patients will be followed until three months after hospital discharge
ICU length of stay | Patients will be followed until ICU discharge, an expected 2 days to 3 weeks.
Weaning Acceleration | Patients will be followed until ICU discharge, an expected 2 days to 3 weeks
Side effects of mobilization protocol | During and 30 minutes after mobilization therapy during ICU stay, approximately 1 to 2 weeks.
  Haemodynamic response to mobilization. Response in systolic and diastolic blood pressure. Response in heart rate. Response in peripheral oxygen saturation.
Length of hospital stay | Patients will be followed until hospital discharge, an expected 4 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Albuquerque, DSc., Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- University Hospital of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Machado ADS, Pires-Neto RC, Carvalho MTX, Soares JC, Cardoso DM, Albuquerque IM. Effects that passive cycling exercise have on muscle strength, duration of mechanical ventilation, and length of hospital stay in critically ill patients: a randomized clinical trial. J Bras Pneumol. 2017 Mar-Apr;43(2):134-139. doi: 10.1590/S1806-37562016000000170. PMID 28538781